CLINICAL TRIAL: NCT00897390
Title: Bioequivalence Study of the Fixed Dose Combination of 2.5 mg Saxagliptin and 1000 mg Metformin Immediate Release (IR) Tablet Relative to 2.5 mg Saxagliptin Tablet and 1000 mg Metformin IR Tablet Co-administered to Healthy Subjects in a Fasted and in a Fed State
Brief Title: Bioequivalence Study of Saxagliptin and Glucophage Combination Formulations in Healthy Subjects (B)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV181-092
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Other): Co-administration of single oral doses of a 2.5 mg tablet of saxagliptin and a 1000 mg tablet of metformin IR under fasted conditions
  Interventions: Drug: Saxagliptin; Drug: Metformin IR (glucophage)
- Arm B (Other): Single oral dose of a FDC tablet consisting of 2.5 mg saxagliptin/ 1000 mg metformin IR under fasted conditions
  Interventions: Drug: Saxagliptin + Metformin IR (FDC)
- Arm C (Other): Co-administration of single oral doses of a 2.5 mg tablet of saxagliptin and a 1000 mg tablet of metformin IR under fed conditions with a standard meal
  Interventions: Drug: Saxagliptin; Drug: Metformin IR (glucophage)
- Arm D (Other): Single oral dose of a FDC tablet consisting of 2.5 mg saxagliptin/ 1000 mg metformin IR under fed conditions with a standard meal
  Interventions: Drug: Saxagliptin + Metformin IR (FDC)

INTERVENTIONS:
Drug: Saxagliptin — Tablet, Oral, 2.5 mg, Once Daily, 1 week
  Other Names: Onglyza
  Arms: Arm A; Arm C
Drug: Metformin IR (glucophage) — Tablets, Oral, 1000 mg, Once Daily, 1 week
  Other Names: Glucophage
  Arms: Arm A; Arm C
Drug: Saxagliptin + Metformin IR (FDC) — Tablet, Oral, Saxagliptin 2.5 mg + metformin IR 1000 mg, Once Daily, 1 Week
  Other Names: Onglyza; Glucophage
  Arms: Arm B; Arm D

SUMMARY:
To demonstrate bioequivalence of a 2.5 mg saxagliptin/1000 mg metformin (glucophage) immediate release (IR) fixed dose combination (FDC) tablet to the 2.5 mg saxagliptin tablet and 1000 mg metformin IR tablet co-administered to healthy subjects in a fasted and in a fed state.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 19 to 45 inclusive
* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m2, inclusive. BMI = weight (kg)/ [height (m)]2

Exclusion Criteria:

* Women of child-bearing potential (WOCBP) who are unwilling or unable to use acceptable barrier methods (condoms and spermicides) to avoid pregnancy for the entire study period and for up to 8 weeks after the last dose of investigational product
* Any significant acute or chronic medical illness
* Current or recent (within 3 months) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* History of allergy to Dipeptidyl peptidase 4 (DPP4) inhibitor or related compounds
* History of allergy or intolerance to metformin or other similar acting agents
* Prior exposure to saxagliptin
* Prior exposure to metformin within 3 months of study drug administration
* Estimated creatinine clearance (Clcr) of < 80ml/min using the Cockcroft Gault formula

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Mds Pharma Services, Lincoln, Nebraska, United States

REFERENCES:
- [Derived] Upreti VV, Keung CF, Boulton DW, Chang M, Li L, Tang A, Hsiang BC, Quamina-Edghill D, Frevert EU, Lacreta FP. Bioequivalence of saxagliptin/metformin immediate release (IR) fixed-dose combination tablets and single-component saxagliptin and metformin IR tablets in healthy adult subjects. Clin Drug Investig. 2013 May;33(5):365-74. doi: 10.1007/s40261-013-0075-z. PMID 23549864
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 58 participants were enrolled in the study; 34 participants were not dosed (23 no longer met study criteria, 4 withdrew consent, and 7 for other reasons).
Groups:
- All Treated Participants: Participants were assigned to 1 of 4 treatment sequences (A-D-B-C, B-A-C-D, C-B-D-A, D-C-A-B). Treatment A=2.5-mg saxagliptin tablet co-administered with 1000-mg metformin IR tablet, fasted; Treatment B=fixed-dose combination (FDC) tablet of 2.5-mg saxagliptin/1000-mg metformin immediate release (IR), fasted; Treatment C=2.5-mg saxagliptin tablet co-administered with 1000-mg metformin IR tablet, fed; Treatment D=FDC tablet of 2.5-mg saxagliptin/1000-mg metformin IR, fed. The washout between each dose was at least 7 days.
Period: Overall Study
Arm/Group | All Treated Participants
Started | 24
Completed | 18
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — No Longer Met Study Criteria | 1
Not completed — Personal Reasons | 1
Not completed — Did not Return for the Clinic Visit | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled and Treated Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20
  Black | 4
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (3.8)
weight [Mean (Standard Deviation); unit: kg] | 79.9 (15.0)

OUTCOME MEASURES:

1. Primary Outcome: Saxagliptin Pharmacokinetic (PK) Parameter Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUC[INF])
Description: Single-dose PK parameters of saxagliptin were derived from plasma concentration versus time data.
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Groups:
- 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted: Co-administration of single oral doses of a 2.5 mg tablet of saxagliptin and a 1000 mg tablet of metformin IR under fasted conditions
- FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted: Single oral dose of a fixed dose combination (FDC) tablet consisting of 2.5 mg saxagliptin/ 1000 mg metformin IR under fasted conditions
- 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed: Co-administration of single oral doses of a 2.5 mg tablet of saxagliptin and a 1000 mg tablet of metformin IR under fed conditions with a standard meal
- FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed: Single oral dose of a FDC tablet consisting of 2.5 mg saxagliptin/ 1000 mg metformin IR under fed conditions with a standard meal
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
ng*h/mL | 47.25 [30.6 to 66.0] | 48.91 [28.7 to 80.7] | 52.89 [37.4 to 75.1] | 51.11 [34.2 to 73.7]
Statistical Analysis 1: Comparison: 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted vs FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted; To demonstrate the bioequivalence of formulation (FDC tablet versus co-administration of separate saxagliptin tablet and metformin IR tablet) in the fasted and fed state, linear mixed model analyses were performed on log(Cmax), log[AUC(INF)] and log[AUC(0-T)] of saxagliptin and metformin, respectively. The factors in the model were sequence, period and treatment as fixed effects and subject within sequence as a random effect; Test type: Non-Inferiority or Equivalence — Point estimates and 90% confidence intervals were calculated for the Arm B to Arm A and Arm D to Arm C ratios of geometric means for Cmax, AUC(INF) and AUC(0-T) of saxagliptin and metformin, respectively. Potency-corrected results were also provided. Bioequivalence will be concluded if the 90% confidence intervals for the test-to-reference ratios of geometric means are entirely contained within 80% to 125% for both Cmax and AUC(INF). No adjustments were made for multiplicity; adjusted geometric mean = 1.042, 90% CI 2-sided [1.009 to 1.075]
Statistical Analysis 2: Comparison: 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed vs FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; adjusted geometric mean = 0.988, 90% CI 2-sided [0.958 to 1.019]

2. Secondary Outcome: BMS-510849 PK Parameter AUC(INF)
Description: Single-dose PK parameters of the active metabolite of saxagliptin, BMS-510849, were derived from plasma concentration versus time data.
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
ng*h/mL | 118.54 [58.7 to 174.4] | 116.19 [48.5 to 212.4] | 127.67 [62.5 to 217.8] | 127.25 [59.4 to 219.3]

3. Primary Outcome: Saxagliptin PK Parameter Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Plasma Concentration (AUC[0-T])
Description: Single-dose PK parameters of saxagliptin were derived from plasma concentration versus time data.
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
ng*h/mL | 44.90 [29.1 to 64.3] | 46.57 [27.8 to 77.7] | 50.50 [35.6 to 73.2] | 49.09 [33.5 to 71.3]
Statistical Analysis 1: Comparison: 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted vs FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; adjusted geometric mean = 1.045, 90% CI 2-sided [1.013 to 1.077]
Statistical Analysis 2: Comparison: 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed vs FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; adjusted geometric mean = 0.992, 90% CI 2-sided [0.962 to 1.022]

4. Primary Outcome: Saxagliptin PK Parameter Maximum Observed Plasma Concentration (Cmax)
Description: Single-dose PK parameters of saxagliptin were derived from plasma concentration versus time data.
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
ng/mL | 8.58 [5.2 to 15.5] | 9.09 [5.5 to 17.1] | 10.97 [7.6 to 18.2] | 10.80 [7.4 to 15.9]
Statistical Analysis 1: Comparison: 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted vs FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; adjusted geometric mean = 1.077, 90% CI 2-sided [0.978 to 1.185]
Statistical Analysis 2: Comparison: 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed vs FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; adjusted geometric mean = 0.987, 90% CI 2-sided [0.900 to 1.083]

5. Primary Outcome: Saxagliptin PK Parameter Plasma Terminal Half-life (T-HALF)
Description: Single-dose PK parameters of saxagliptin were derived from plasma concentration versus time data.
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
hours | 6.66 (1.185) | 6.34 (0.941) | 6.47 (1.529) | 5.78 (1.333)

6. Primary Outcome: Saxagliptin PK Parameter Time of Maximum Observed Plasma Concentration (Tmax)
Description: Single-dose PK parameters of saxagliptin were derived from plasma concentration versus time data.
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Median (Full Range); unit: hours
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
hours | 1.50 [0.5 to 4.0] | 0.75 [0.3 to 3.0] | 1.00 [0.3 to 3.0] | 1.50 [0.3 to 3.0]

7. Primary Outcome: Metformin PK Parameter AUC(INF)
Description: Single-dose PK parameters of metformin were derived from plasma concentration versus time data.
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
ng*h/mL | 13363.46 [8872.9 to 19164.2] | 12677.92 [8827.3 to 16811.6] | 12357.87 [6875.3 to 15926.2] | 12126.19 [7328.6 to 15424.7]
Statistical Analysis 1: Comparison: 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted vs FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; adjusted geometric mean = 0.974, 90% CI 2-sided [0.921 to 1.030]
Statistical Analysis 2: Comparison: 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed vs FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; adjusted geometric mean = 0.966, 90% CI [0.915 to 1.020]

8. Primary Outcome: Metformin PK Parameter AUC(0-T)
Description: Single-dose PK parameters of metformin were derived from plasma concentration versus time data.
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
ng*h/mL | 13238.43 [8782.0 to 18991.8] | 12400.41 [8105.3 to 16603.8] | 12124.31 [6629.2 to 15842.4] | 11996.88 [7142.5 to 15326.6]
Statistical Analysis 1: Comparison: 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted vs FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; adjusted geometric mean = 0.962, 90% CI [0.906 to 1.020]
Statistical Analysis 2: Comparison: 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed vs FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; adjusted geometric mean = 0.974, 90% CI [0.920 to 1.032]

9. Primary Outcome: Metformin PK Parameter Cmax
Description: Single-dose PK parameters of metformin were derived from plasma concentration versus time data.
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
ng/mL | 2004.99 [1187.2 to 3144.6] | 1830.76 [1142.5 to 2662.5] | 1666.55 [768.7 to 2256.5] | 1642.90 [848.1 to 2018.3]
Statistical Analysis 1: Comparison: 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted vs FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; adjusted geometric mean = 0.937, 90% CI 2-sided [0.864 to 1.016]
Statistical Analysis 2: Comparison: 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed vs FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; adjusted geometric mean = 0.964, 90% CI 2-sided [0.891 to 1.042]

10. Primary Outcome: Metformin PK Parameter T-HALF
Description: Single-dose PK parameters of metformin were derived from plasma concentration versus time data.
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
hours | 8.43 (2.956) | 10.58 (8.895) | 11.78 (5.999) | 7.63 (2.309)

11. Primary Outcome: Metformin PK Parameter Tmax
Description: Single-dose PK parameters of metformin were derived from plasma concentration versus time data.
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Median (Full Range); unit: hours
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
hours | 2.00 [1.0 to 4.0] | 2.98 [1.5 to 4.0] | 4.00 [2.0 to 4.0] | 4.00 [3.0 to 4.0]

12. Secondary Outcome: BMS-510849 PK Parameter AUC(0-T)
Description: as for outcome 2
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
ng*h/mL | 108.31 [52.0 to 169.2] | 106.11 [42.3 to 201.4] | 117.42 [54.3 to 210.7] | 117.43 [51.1 to 210.9]

13. Secondary Outcome: BMS-510849 PK Parameter Cmax
Description: as for outcome 2
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
ng/mL | 16.77 [6.4 to 32.8] | 15.17 [4.7 to 32.0] | 18.24 [7.6 to 36.5] | 18.58 [6.2 to 33.5]

14. Secondary Outcome: BMS-510849 PK Parameter T-Half
Description: Single-dose PK parameters of the active metabolite of saxagliptin, BMS-510849, were derived from their respective plasma concentration versus time data.
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
hours | 8.05 (1.427) | 7.31 (1.369) | 7.48 (1.504) | 7.35 (1.622)

15. Secondary Outcome: BMS-510849 PK Parameter T-Max
Description: as for outcome 2
Time Frame: pre-dose, post-dose at 15, 30, 45, 90 minutes, hours 1, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 of each period
Population: Treated participants with PK measures
Measure: Median (Full Range); unit: hours
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
hours | 2.00 [1.0 to 4.0] | 2.00 [0.8 to 4.0] | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]

16. Secondary Outcome: Deaths, Serious Adverse Events (SAEs), Adverse Events (AEs), and Discontinuations Due to AEs
Description: An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a patient or clinical investigation subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: AEs collected from Day 1/Period 1 through study discharge (study duration: approximately 45 days). SAEs collected from date of written consent until 30 days post discontinuation of dosing or subject's participation in the study.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
participants
  Deaths | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 0 | 0
  AEs | 5 | 2 | 4 | 3
  Discontinuations dues to AEs | 0 | 0 | 1 | 1

17. Secondary Outcome: AEs of Special Interest
Description: See Outcome Measure 16 for a definition of AEs. AEs of clinical interest for saxagliptin were defined as those relating to the following:skin disorders, infection-related AEs (system organ class [SOC]: Infections and Infestations), thrombocytopenia, lymphopenia, hypoglycemia, cardiovascular AEs indicative of acute cardiovascular events, localized edema, fractures, pancreatitis, and AEs of hypersensitivity.
Time Frame: AEs collected from Day 1/Period 1 through study discharge (study duration: approximately 45 days).
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 21 | 22
participants | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities (MA)
Description: Laboratory abnormalities=any result that is clinically significant, met the definition of an SAE, required discontinuation or interruption of study drug, or required specific corrective therapy. Upper normal (UN)/lower normal (LN) values: leukocytes UN, 11.40x10^3 c/uL; absolute neutrophils/bands LN, 1.500x10^3 c/uL; aspartate aminotransferase UN, 48 U/L; alanine aminotransferase UN, 67 U/L; blood urea nitrogen UN, 20.0 mg/dL; creatine kinase UN, 350 U/L; lactate dehydrogenase UN, 249 U/L.
Time Frame: Within 21 days of study Day 1, Days 1-3 of Periods 1, 2, 3, and 4.
Population: Treated participants. One participant each in Arm C and Arm D was not evaluated for this measure.
Measure: Number; unit: participants
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 20 | 21
participants
  Leukocytes - High(>1.2 * upper limit normal [ULN]) | 0 | 0 | 0 | 1
  Abs. Neutrophils/Bands-Low (<=lower LN [LLN]) | 1 | 1 | 1 | 1
  Aspartate Aminotransferase - High (>1.25 * ULN) | 0 | 0 | 0 | 1
  Alanine Aminotransferase - High (>1.25 * ULN) | 0 | 0 | 0 | 1
  Blood Urea Nitrogen - High (1.1 * ULN) | 0 | 1 | 1 | 0
  Creatine Kinase - High (>1.5 ULN) | 1 | 1 | 0 | 2
  Lactate Dehydrogenase - High (>1.25 ULN) | 0 | 0 | 0 | 1

19. Secondary Outcome: Number of Participants With Marked Urinalysis Abnormalities
Description: Protein, Urine Abnormality: if value >= 2+ (or if pretreatment value >= 1+, then >= 2 * pretreatment). Glucose, Urine Abnormality: if value >= 2+ (or if pretreatment value >= 1+, then >= 2 * pretreatment). Blood, Urine Abnormality: if value >= 2+ (or if pretreatment value >= 1+, then >= 2 * pretreatment). White Blood Cell (WBC), Urine Abnormality: if value >= 2+ (or if pretreatment value >= 2+, then >= 4+). Red Blood Cell (RBC), Urine Abnormality: if value >= 2+ (or if pretreatment value >= 2+, then >= 4+). (The '+' is a normal lab result and refers to the magnitude of the finding.)
Time Frame: Within 21 days of study Day 1, Days 1-3 of Periods 1, 2, 3, and 4.
Population: Number of Participants Analyzed=treated participants; n=number of participants evaluated for this measure (among the 6 participants who had the urinary WBC and RBC test, there are only 2 had a pre-study evaluation, and were therefore evaluable for these measures.
Measure: Number; unit: participants
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 20 | 21
participants
  Protein, Urine (n=19, 19, 20, 21) | 0 | 0 | 0 | 0
  Glucose, Urine (n=19, 19, 20, 21) | 0 | 0 | 0 | 0
  Blood, Urine (n=19, 19, 20, 21) | 1 | 0 | 0 | 2
  White Blood Cells, Urine (n=2, 2, 2, 2) | 0 | 0 | 1 | 0
  Red Blood Cells, Urine (n=2, 2, 2, 2) | 0 | 0 | 0 | 0

20. Secondary Outcome: Electrocardiogram (ECG), Vital Sign, and Physical Finding Abnormalities
Description: 12-lead Electrocardiogram (ECG), Vital Sign (body temperature, respiratory rate, seated blood pressure and heart rate), and Physical Finding Abnormalities reported by investigator as AEs.
Time Frame: At Screening (within 21 days of Study Day 1), Day -1 of Period 1 (ECG and Physical only), Day 1 of Periods 1-4 (Vitals only), at Study Discharge (Day 3 of Period 4) or Discontinuation
Population: Treated participants. One participant each in Arm C and Arm D was not evaluated for this measure.
Measure: Number; unit: participants
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed
Number analyzed (Participants) | 19 | 19 | 20 | 21
participants
  ECG Abnormalities | 0 | 0 | 0 | 0
  Vital Sign Abnormalities | 0 | 0 | 0 | 0
  Physical Finding Abnormalities | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted: Single oral dose of a FDC tablet consisting of 2.5 mg saxagliptin/ 1000 mg metformin IR under fasted conditions
- Not Dosed: 58 participants were enrolled in the study; 34 participants were not dosed (23 no longer met study criteria, 4 withdrew consent, and 7 for other reasons).
Arm/Group | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed | Not Dosed
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/21 | 0/24 | 0/34
Other Adverse Events (participants affected / at risk) | 3/19 | 2/19 | 2/21 | 3/24 | 0/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fasted (N=19) | FDC Tablet 2.5-mg Saxa/1000-mg Met Tablet, Fasted (N=19) | 2.5-mg Saxa Tablet/1000-mg Met Tablet, Fed (N=21) | FDC Tablet of 2.5-mg Saxa/1000-mg Met Tablet, Fed (N=24) | Not Dosed (N=34)
EYE DISCHARGE (Eye disorders) | 0/6 | 0/6 | 1/6 | 0/6 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1/6 | 0/6 | 0/6 | 0/6 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1/6 | 0/6 | 0/6 | 0/6 | 0
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1/6 | 0/6 | 0/6 | 0/6 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1/6 | 0/6 | 0/6 | 0/6 | 0
PALPITATIONS (Cardiac disorders) | 0/6 | 1/6 | 0/6 | 0/6 | 0
HEADACHE (Nervous system disorders) | 1/6 | 2/6 | 2/6 | 1/6 | 0
DIZZINESS (Nervous system disorders) | 0/6 | 1/6 | 0/6 | 0/6 | 0
NAUSEA (Gastrointestinal disorders) | 1/6 | 0/6 | 1/6 | 0/6 | 0
VOMITING (Gastrointestinal disorders) | 1/6 | 0/6 | 0/6 | 0/6 | 0
DIARRHOEA (Gastrointestinal disorders) | 0/6 | 0/6 | 1/6 | 2/6 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0/6 | 0/6 | 1/6 | 0/6 | 0
FLATULENCE (Gastrointestinal disorders) | 0/6 | 0/6 | 1/6 | 1/6 | 0
CONSTIPATION (Gastrointestinal disorders) | 0/6 | 0/6 | 1/6 | 0/6 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0/6 | 0/6 | 0/6 | 1/6 | 0
EAR PAIN (Ear and labyrinth disorders) | 0/6 | 0/6 | 1/6 | 1/6 | 0
EAR DISCOMFORT (Ear and labyrinth disorders) | 1/6 | 0/6 | 0/6 | 0/6 | 0
MENSTRUATION DELAYED (Reproductive system and breast disorders) | 0/6 | 1/6 | 0/6 | 0/6 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1/6 | 0/6 | 0/6 | 0/6 | 0
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0/6 | 0/6 | 1/6 | 0/6 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1/6 | 0/6 | 0/6 | 0/6 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1/6 | 0/6 | 0/6 | 0/6 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0/6 | 0/6 | 1/6 | 0/6 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1/6 | 0/6 | 0/6 | 0/6 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0/6 | 0/6 | 1/6 | 1/6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.